CLINICAL TRIAL: NCT06585852
Title: Efficacy of Xenograft Alone or Mixed With Arginyl-Glycyl-Aspartic Acid (RGD) in Horizontal Ridge Augmentation With Split-crest Technique for Implant Placement. A Randomized Clinical Trial
Brief Title: Efficacy of Xenograft Alone or Mixed With Arginyl-Glycyl-Aspartic Acid (RGD) in Horizontal Ridge Augmentation With Split-crest Technique for Implant Placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, muhammed nagy, Principle investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RGD in Ridge splitting
Record Dates: First submitted 2024-09-01; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Implant Dentistry
MeSH Terms: interventions — Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Xenograft alone with split-crest technique by ultrasonic bone surgery and implant placement.
  Interventions: Drug: Xenograft; Procedure: Split crest technique
- Study Group (Experimental): Xenograft mixed with RGD with split-crest technique by ultrasonic bone surgery and implant placement.
  Interventions: Drug: RGD; Drug: Xenograft; Procedure: Split crest technique

INTERVENTIONS:
Drug: RGD — Study group main material
  Other Names: Arginylglycylaspartic acid
  Arms: Study Group
Drug: Xenograft — Scaffold material of choice
Procedure: Split crest technique — Piezoelectric surgery

SUMMARY:
The aim of the present study is to evaluate the efficacy of xenograft alone or xenograft mixed with Arginylglycylaspartic acid (RGD) , in horizontal ridge augmentation with split-crest technique, for implant placement.

DETAILED DESCRIPTION:
A comparative study for ridge augmentation procedure, With two groups. First group underwent a surgical ridge splitting procedure with ultrasonic bone surgery and grafting with Xenograft alone and implant placement. Second group underwent a surgical ridge splitting procedure with ultrasonic bone surgery Xenograft mix ed with Arginylglycylaspartic acid (RGD) and implant placement.

Both groups were followed up for 1 and 3 months after loading.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age 18-30) exhibiting initial insufficiently bone width.
2. Patients with good oral hygiene.
3. Patients must be free from systemic diseases that may influence the outcome of the therapy.
4. Patients with bony horizontal defects alone, Class III & IV.

Exclusion Criteria:

1. Heavy smokers.
2. Patient treated by immunosuppressive chemotherapy or radio therapy,
3. Allergy to any material or medication used in the study.
4. Pregnant females.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
ISQ measurement for implant stability | At time of surgery, at loading and 3 months after loading.
  Evaluate implant stability by osstell device

SECONDARY OUTCOMES:
Bone density around dental implants. | At time of loading and 3 months after loading
  Evaluation of bone density after ridge splitting and implant placement

CONTACTS AND LOCATIONS:
Locations (1):
- Al Azhar University of Cairo, Cairo, Nasr City, Egypt